CLINICAL TRIAL: NCT04039919
Title: A Double-Blind, Placebo-Controlled, Randomized, Single-Center, Cross-Over Study to Investigate the Pharmacodynamic, Pharmacokinetic, Safety, and Tolerability Profiles of Padsevonil in Healthy Study Participants Receiving Either Ethanol or Cannabidiol
Brief Title: A Study to Test the Pharmacodynamic, Pharmacokinetic, Safety, and Tolerability of Padsevonil in Healthy Study Participants Receiving Either Ethanol or Cannabidiol
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizures
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0071; 2019-000703-32 (EudraCT Number)
Record Dates: First submitted 2019-07-12; First posted 2019-07-31 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Healthy Participants
Keywords: Ethanol; Cannabidiol; Padsevonil
MeSH Terms: interventions — padsevonil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: Padsevonil and Ethanol (Experimental): Subjects will be randomized to receive Padsevonil and Ethanol.
  Interventions: Drug: Padsevonil
- Part A: Padsevonil and Ethanol-Placebo (Placebo Comparator): Subjects will be randomized to receive Padsevonil and Ethanol-Placebo.
  Interventions: Drug: Padsevonil
- Part A: Ethanol and Ethanol-Placebo (No Intervention): Subjects will be randomized to receive Ethanol and Ethanol-Placebo.
- Part A: Ethanol-Placebo and Ethanol (No Intervention): Subjects will be randomized to receive Ethanol and Ethanol-Placebo.
- Part B: Padsevonil and Cannabidiol (Experimental): Subjects will be randomized to receive Padsevonil and Cannabidiol.
  Interventions: Drug: Padsevonil
- Part B: Padsevonil-Placebo and Cannabidiol (Placebo Comparator): Subjects will be randomized to receive Padsevonil-Placebo and Cannabidiol.
  Interventions: Drug: Placebo (PSL)

INTERVENTIONS:
Drug: Padsevonil — Padsevonil will be administered in predefined dosages.
  Arms: Part A: Padsevonil and Ethanol; Part A: Padsevonil and Ethanol-Placebo; Part B: Padsevonil and Cannabidiol
Drug: Placebo (PSL) — Placebo will be provided matching Padsevonil to maintain the blinding.
  Arms: Part B: Padsevonil-Placebo and Cannabidiol

SUMMARY:
The purpose of the study is to evaluate the pharmacodynamic (PD) interaction between steady-steady treatment with padsevonil (PSL) and Ethanol and the pharmacokinetic (PK) interaction between stead-state treatment with PSL and cannabidiol (CBD).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participant must have previous experience with alcohol consumption and, therefore, must be familiar with the effects and able to tolerate social amounts of alcohol
* Participant has a body weight of at least 50 kg (males) or 45 kg (females) and body mass index (BMI) within the range 18 to 30 kg/m2 (inclusive)
* Participants are male or female:
* A male participant must agree to use contraception as detailed in the protocol during the treatment period and for at least 7 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:
* Not a woman of childbearing potential (WOCBP) as defined n the protocol OR
* A WOCBP who agrees to follow the contraceptive guidance in the protocol during the Treatment Period and for at least 90 days after the last dose of study treatment

Exclusion Criteria:

* Participant has history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Participant has a history of chronic alcohol or drug abuse within the previous 6 months or the presence of drug or alcohol dependency at Screening or Day -1 or tests positive for alcohol and/or drugs at Screening or Day -1
* Participant has a known hypersensitivity to any components of the study medication or comparative drugs (and/or an investigational device) as stated in this protocol
* Participant has a history of unexplained syncope or a family history of sudden death due to long QT syndrome
* Participant has lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Participant has past or intended use of over-the-counter or prescription medication including herbal medications within 2 weeks or 5 half-lives prior to dosing
* Participant has used hepatic enzyme-inducing drugs within 2 months prior to dosing
* Participant has alanine transaminase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN)
* Participant has current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Participant has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline
* Participant has the presence of hepatitis B surface antigen (HBsAg) at Screening or within 3 months prior to dosing
* Participant has a positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention
* Participant has a positive human immunodeficiency virus (HIV) antibody test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0071 001, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in July 2019 and concluded in May 2020.
Pre-assignment Details: Participant Flow refers to the All Study Participants Set which included all participants who have signed the Informed Consent form (ICF).
Groups:
- Part A: Treatment Sequence A: Participants received ethanol 0.6 grams per liter (g/L) intravenous (IV) infusion on Day 1 during Treatment Period 1 (TP1), followed by placebo (for ethanol IV infusion) on Day 1 during TP2, then padsevonil (PSL) oral tablets 100 mg or 200 mg BID on Day 1 to 4 during TP3, PSL 200 mg BID oral tablets + Ethanol IV infusion on Day 5 during TP4, PSL oral tablets 100 mg or 200 mg + Placebo (for ethanol IV infusion) on Day 7 during TP5, and then PSL 100 mg BID oral tablets on Day 9 during TP6. There was a washout of at least 2 days between Treatment Periods 2 and 3.
- Part A: Treatment Sequence B: Participants received ethanol 0.6 g/L IV infusion on Day 1 during TP1, followed by placebo (for ethanol IV infusion) on Day 1 during TP2, then PSL oral tablets 100 mg or 200 mg BID on Day 1 to 4 during TP3, PSL oral tablets 100 mg or 200 mg + Placebo (for ethanol IV infusion) on Day 5 during TP4, PSL 200 mg BID oral tablets + Ethanol IV infusion on Day 7 during TP5, and then PSL 100 mg BID oral tablets on Day 9 during TP6. There was a washout of at least 2 days between Treatment Periods 2 and 3.
- Part A: Treatment Sequence C: Participants received placebo (for ethanol IV infusion) on Day 1 during TP1, followed by ethanol 0.6 g/L IV infusion on Day 1 during TP2, then PSL oral tablets 100 mg or 200 mg BID on Day 1 to 4 during TP3, PSL 200 mg BID oral tablets + Ethanol IV infusion on Day 5 during TP4, PSL oral tablets 100 mg or 200 mg + Placebo (for ethanol IV infusion) on Day 7 during TP5, and then PSL 100 mg BID oral tablets on Day 9 during TP6. There was a washout of at least 2 days between Treatment Periods 2 and 3.
- Part A: Treatment Sequence D: Participants received placebo (for ethanol IV infusion) on Day 1 during TP1, followed by ethanol 0.6 g/L IV infusion on Day 1 during TP2, then PSL oral tablets 100 mg or 200 mg BID on Day 1 to 4 during TP3, PSL oral tablets 100 mg or 200 mg + Placebo (for ethanol IV infusion) on Day 5 during TP4, PSL 200 mg BID oral tablets + Ethanol IV infusion on Day 7 during TP5, and then PSL 100 mg BID oral tablets on Day 9 during TP6. There was a washout of at least 2 days between Treatment Periods 2 and 3.
- Part B: Cannabidiol (CBD): Participants received a single oral dose of CBD 10 milligrams per kilogram (mg/kg) solution, under fasted condition on Day 1 during TP1.
Period: Treatment Period 1
Arm/Group | Part A: Treatment Sequence A | Part A: Treatment Sequence B | Part A: Treatment Sequence C | Part A: Treatment Sequence D | Part B: Cannabidiol (CBD)
Started | 7 | 6 | 5 | 6 | 16
Completed | 6 | 6 | 5 | 6 | 0
Not Completed | 1 | 0 | 0 | 0 | 16
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor's decision | 0 | 0 | 0 | 0 | 16
Period: Treatment Period 2
Arm/Group | Part A: Treatment Sequence A | Part A: Treatment Sequence B | Part A: Treatment Sequence C | Part A: Treatment Sequence D | Part B: Cannabidiol (CBD)
Started | 6 | 6 | 5 | 6 | 0
Completed | 6 | 6 | 5 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Part A: Treatment Sequence A | Part A: Treatment Sequence B | Part A: Treatment Sequence C | Part A: Treatment Sequence D | Part B: Cannabidiol (CBD)
Started | 6 | 6 | 5 | 6 | 0
Completed | 6 | 6 | 5 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Part A: Treatment Sequence A | Part A: Treatment Sequence B | Part A: Treatment Sequence C | Part A: Treatment Sequence D | Part B: Cannabidiol (CBD)
Started | 6 | 6 | 5 | 6 | 0
Completed | 6 | 6 | 5 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | Part A: Treatment Sequence A | Part A: Treatment Sequence B | Part A: Treatment Sequence C | Part A: Treatment Sequence D | Part B: Cannabidiol (CBD)
Started | 6 | 6 | 5 | 6 | 0
Completed | 5 | 6 | 5 | 6 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 6
Arm/Group | Part A: Treatment Sequence A | Part A: Treatment Sequence B | Part A: Treatment Sequence C | Part A: Treatment Sequence D | Part B: Cannabidiol (CBD)
Started | 5 | 6 | 5 | 6 | 0
Completed | 5 | 6 | 5 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Safety Set (SS) which consisted of all study participants who were randomized and had received at least 1 dose (any amount) of study medication.
Arm/Group | Part A: Treatment Sequence A | Part A: Treatment Sequence B | Part A: Treatment Sequence C | Part A: Treatment Sequence D | Part B: Cannabidiol (CBD) | Total Title
Number analyzed (Participants) | 7 | 6 | 5 | 6 | 16 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 5 | 6 | 16 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (9.9) | 30.8 (9.1) | 28.4 (7.0) | 30.7 (4.1) | 27.9 (9.3) | 29.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 1 | 11 | 18
  Male | 6 | 2 | 4 | 5 | 5 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 5 | 5 | 4 | 15 | 36
  Other or Mixed | 0 | 1 | 0 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Smooth Pursuit Eye Movements on Day 1 of Period 1 or Day 3 of Period 2 During Part A
Description: Smooth pursuit to assess eye movement coordination and attention to evaluate the ethanol effect. The average percentage of smooth pursuit for all stimulus frequencies was used as a parameter. Participants received either ethanol or placebo on Day 1 of Period 1 or on Day 3 of Period 2. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours postdose on Day 1 of Period 1 or Day 3 of Period 2
Population: Full Analysis Set (FAS) consisted of all study participants that were randomized, received study medication, and had at least one valid post-baseline primary pharmacodynamic assessment observation. Here, n (number analyzed) signifies participants evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: percentage of eye movements
Groups:
- Part A: Ethanol (FAS): Participants received ethanol 0.6 g/L IV infusion on Day 1 during TP1 in Treatment Sequence A and B and on Day 1 during TP2 in Treatment Sequence C and D. Participants formed the FAS.
- Part A: Placebo (FAS): Participants received matching placebo (for ethanol IV infusion) on Day 1 during TP1 in Treatment Sequence A and B and on Day 1 during TP2 in Treatment Sequence C and D. Participants formed the Full Analysis Set (FAS).
Arm/Group | Part A: Ethanol (FAS) | Part A: Placebo (FAS)
Number analyzed (Participants) | 24 | 23
percentage of eye movements
  Predose | 44.838 (9.110) | 43.252 (8.688)
  0.5 hour | 38.046 (8.674) | 43.661 (9.345)
  1 hour | 37.604 (8.574) | 43.748 (10.298)
  2 hours | 37.300 (8.778) | 42.930 (9.636)
  3 hours: number analyzed (Participants) | 23 | 23
  3 hours | 36.726 (7.441) | 42.809 (10.639)
  4 hours: number analyzed (Participants) | 23 | 23
  4 hours | 36.822 (8.405) | 42.478 (9.351)
  5 hours: number analyzed (Participants) | 23 | 23
  5 hours | 35.913 (7.359) | 42.622 (9.200)
  6 hours: number analyzed (Participants) | 23 | 23
  6 hours | 40.570 (9.353) | 43.300 (8.960)
  8 hours: number analyzed (Participants) | 23 | 23
  8 hours | 41.948 (10.245) | 44.026 (10.085)
  10 hours: number analyzed (Participants) | 23 | 23
  10 hours | 43.491 (8.928) | 43.504 (11.394)

2. Primary Outcome: Percentage of Smooth Pursuit Eye Movements on Day 5 of Period 4 or Day 7 of Period 5 During Part A
Description: Smooth pursuit to assess eye movement coordination and attention to evaluate the ethanol effect. The average percentage of smooth pursuit for all stimulus frequencies was used as a parameter. Participants received either ethanol or placebo on Day 5 of Period 4 or Day 7 of Period 5. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours postdose on Day 5 of Period 4 or Day 7 of Period 5
Population: FAS consisted of all study participants that were randomized, received study medication, and had at least one valid post-baseline primary pharmacodynamic assessment observation. Here, Number of participants analyzed signifies participants who were evaluable for the assessment.
Measure: Mean (Standard Deviation); unit: percentage of eye movements
Groups:
- Part A: PSL + Ethanol (FAS): Participants received PSL 200 mg BID oral tablets + Ethanol IV infusion on Day 5 during TP4 in Treatment Sequence A and C and on Day 7 during TP5 in Treatment Sequence B and D. Participants formed the FAS.
- Part A: PSL + Placebo (FAS): Participants received PSL oral tablets 100 mg or 200 mg + Placebo (for ethanol IV infusion) on Day 7 during TP5 in Treatment Sequence A and C and on Day 5 during TP4 in Treatment Sequence B and D. Participants formed the FAS.
Arm/Group | Part A: PSL + Ethanol (FAS) | Part A: PSL + Placebo (FAS)
Number analyzed (Participants) | 23 | 22
percentage of eye movements
  Predose | 41.107 (9.930) | 41.402 (8.500)
  0.5 hour | 32.591 (7.140) | 39.655 (9.703)
  1 hour | 30.874 (6.790) | 35.814 (7.893)
  2 hours | 28.309 (5.321) | 36.036 (9.172)
  3 hours | 28.530 (6.881) | 36.727 (9.512)
  4 hours | 30.400 (9.466) | 36.668 (8.411)
  5 hours | 30.239 (6.750) | 35.714 (8.865)
  6 hours | 33.761 (8.383) | 38.945 (9.676)
  8 hours | 35.604 (8.894) | 37.973 (8.849)
  10 hours | 38.570 (10.683) | 38.591 (9.508)

3. Primary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of Padsevonil During Part B
Description: Cmax is maximum observed plasma concentration at steady state of padsevonil.
Time Frame: Predose up to 12 hours postdose
Population: Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.
Groups:
- Part B: PSL: Zero participants received PSL during Part B because the study was terminated.
Arm/Group | Part B: PSL
Number analyzed (Participants) | 0

4. Primary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of Cannabidiol During Part B
Description: Cmax is maximum observed plasma concentration at steady state of CBD.
Time Frame: Predose up to 12 hours postdose
Population: Pharmacokinetic Set (PKS) included all study participants that received at least one dose of active study drug and have at least one observable pharmacokinetic measurement.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter
Groups:
- Part B: CBD (PKS): Participants received a single oral dose of CBD 10 mg/kg solution, under fasted condition on Day 1 during TP1. Participants formed the PKS.
Arm/Group | Part B: CBD (PKS)
Number analyzed (Participants) | 16
nanograms per milliliter | NA [NA to NA] — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

5. Primary Outcome: Area Under the Curve Over a Dosing Interval (AUCtau) of Padsevonil During Part B
Description: AUCtau is the area under the curve over a dosing interval of padsevonil.
Time Frame: Predose up to 12 hours post dose
Population: as for outcome 3
Arm/Group | Part B: PSL
Number analyzed (Participants) | 0

6. Primary Outcome: Area Under the Curve Over a Dosing Interval (AUCtau) of Cannabidiol During Part B
Description: AUCtau is the area under the curve over a dosing interval of CBD.
Time Frame: Predose up to 12 hours postdose
Population: PKS included all study participants that received at least one dose of active study drug and have at least one observable pharmacokinetic measurement.
Measure: Geometric Mean (95% Confidence Interval); unit: hours*nanogram per milliliter
Arm/Group | Part B: CBD (PKS)
Number analyzed (Participants) | 16
hours*nanogram per milliliter | NA [NA to NA] — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

7. Secondary Outcome: Breath Concentration of Ethanol Over Time on Day 1 of Period 1 or Day 3 of Period 2 During Part A
Description: Continuous infusion of ethanol began with a 30 minute loading phase (prior to 0 hours) and was continued for 5 hours with adjustments during the infusion. Participants received either ethanol on Day 1 of Period 1 or on Day 3 of Period 2. Therefore, the results were summarized by treatment.
Time Frame: -0.4, -0.3, -0.2, -0.16, -0.08, Predose, 0.16, 0.3, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7 and 8 hours postdose on Day 1 of Period 1 or on Day 3 of Period 2
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: grams per liter
Groups:
- Part A: Ethanol (PKS): Participants received ethanol 0.6 g/L IV infusion on Day 1 during TP1 in Treatment Sequence A and B and on Day 1 during TP2 in Treatment Sequence C and D. Participants formed the Pharmacokinetic Set (PKS).
Arm/Group | Part A: Ethanol (PKS)
Number analyzed (Participants) | 21
grams per liter
  -0.4 hour | 0.290 [0.254 to 0.333]
  -0.3 hour | 0.428 [0.379 to 0.483]
  -0.2 hour | 0.477 [0.446 to 0.511]
  -0.16 hour | 0.530 [0.499 to 0.564]
  -0.08 hour | 0.562 [0.539 to 0.585]
  Predose | 0.555 [0.538 to 0.571]
  0.16 hour | 0.578 [0.558 to 0.599]
  0.3 hour | 0.592 [0.574 to 0.611]
  0.5 hour | 0.574 [0.552 to 0.598]
  1 hour | 0.552 [0.525 to 0.581]
  1.5 hours | 0.557 [0.533 to 0.583]
  2 hours | 0.568 [0.544 to 0.593]
  2.5 hours | 0.574 [0.547 to 0.601]
  3 hours | 0.572 [0.544 to 0.602]
  3.5 hours | 0.574 [0.556 to 0.593]
  4 hours | 0.593 [0.575 to 0.612]
  4.5 hours | 0.603 [0.583 to 0.624]
  5 hours | 0.590 [0.575 to 0.605]
  6 hours | 0.356 [0.322 to 0.394]
  7 hours | 0.172 [0.139 to 0.213]
  8 hours | 0.105 [0.073 to 0.151]

8. Secondary Outcome: Breath Concentration of Ethanol Over Time on Day 5 of Period 4 or Day 7 of Period 5 During Part A
Description: Continuous infusion of ethanol began with a 30 minute loading phase (prior to 0 hours) and was continued for 5 hours with adjustments during the infusion. Participants received either ethanol on Day 5 of Period 4 or Day 7 of Period 5. Therefore, the results were summarized by treatment.
Time Frame: -0.4, -0.3, -0.2, -0.16, -0.08, Predose, 0.16, 0.3, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7 and 8 hours postdose on Day 5 of Period 4 or Day 7 of Period 5
Population: PKS included all study participants that received at least one dose of active study drug and have at least one observable pharmacokinetic measurement. Here, n (number analyzed) signifies participants evaluable at specified time points only.
Measure: Geometric Mean (95% Confidence Interval); unit: grams per liter
Groups:
- Part A: PSL + Ethanol (PKS): Participants received PSL 200 mg BID oral tablets + Ethanol IV infusion on Day 5 during TP4 in Treatment Sequence A and C and on Day 7 during TP5 in Treatment Sequence B and D. Participants formed the PKS.
Arm/Group | Part A: PSL + Ethanol (PKS)
Number analyzed (Participants) | 21
grams per liter
  -0.4 hour | 0.321 [0.281 to 0.367]
  -0.3 hour | 0.464 [0.417 to 0.516]
  -0.2 hour | 0.499 [0.451 to 0.553]
  -0.16 hour | 0.524 [0.492 to 0.558]
  -0.08 hour | 0.505 [0.468 to 0.545]
  Predose | 0.499 [0.467 to 0.533]
  0.16 hour | 0.591 [0.567 to 0.617]
  0.3 hour | 0.622 [0.606 to 0.639]
  0.5 hour | 0.608 [0.591 to 0.624]
  1 hour | 0.581 [0.560 to 0.603]
  1.5 hours | 0.566 [0.544 to 0.588]
  2 hours | 0.566 [0.540 to 0.593]
  2.5 hours | 0.579 [0.550 to 0.608]
  3 hours | 0.608 [0.585 to 0.631]
  3.5 hours | 0.602 [0.582 to 0.623]
  4 hours | 0.612 [0.593 to 0.632]
  4.5 hours | 0.610 [0.590 to 0.631]
  5 hours | 0.613 [0.590 to 0.637]
  6 hours | 0.373 [0.338 to 0.411]
  7 hours: number analyzed (Participants) | 20
  7 hours | 0.199 [0.171 to 0.232]
  8 hours | 0.084 [0.066 to 0.108]

9. Secondary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of Padsevonil During Part A
Description: Cmax,ss is the maximum observed plasma concentration at steady state of padsevonil.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 12 hours postdose on Day 5
Population: PKS included all study participants that received at least one dose of active study drug and have at least one observable pharmacokinetic measurement. Here, Number of participants analyzed signifies participants who were evaluable for the assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter
Groups:
- Part A: PSL + Placebo (PKS): Participants received PSL oral tablets 100 mg or 200 mg + Placebo (for ethanol IV infusion) on Day 7 during TP5 in Treatment Sequence A and C and on Day 5 during TP4 in Treatment Sequence B and D. Participants formed the PKS.
Arm/Group | Part A: PSL + Ethanol (PKS) | Part A: PSL + Placebo (PKS)
Number analyzed (Participants) | 20 | 21
nanograms per milliliter | 832.9 [488.3 to 1421] | 1077 [778.6 to 1489]
Statistical Analysis 1: Comparison: Part A: PSL + Ethanol (PKS) vs Part A: PSL + Placebo (PKS); The log-transformed PK parameters was analyzed by a mixed analysis of variance (ANOVA) with period and treatment as fixed effects and study participant as the random effect. The estimates and confidence intervals are back-transformed after the analysis; Test type: Other; Geometric LS Mean ratio = 0.7850, 90% CI 2-sided [0.6513 to 0.9461]

10. Secondary Outcome: Area Under the Curve Over a Dosing Interval (AUCtau) of Padsevonil During Part A
Description: AUC0-tau is the area under the curve over a dosing interval of padsevonil.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 12 hours postdose on Day 5
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: hours*nanogram per milliliter
Arm/Group | Part A: PSL + Ethanol (PKS) | Part A: PSL + Placebo (PKS)
Number analyzed (Participants) | 20 | 20
hours*nanogram per milliliter | 3504 [2010 to 6109] | 4289 [2904 to 6335]
Statistical Analysis 1: Comparison: Part A: PSL + Ethanol (PKS) vs Part A: PSL + Placebo (PKS); The log-transformed PK parameters was analyzed by a mixed ANOVA with period and treatment as fixed effects and study participant as the random effect. The estimates and confidence intervals are back-transformed after the analysis; Test type: Other; Geometric LS Mean Ratio = 0.8342, 90% CI 2-sided [0.6999 to 0.9942]

11. Secondary Outcome: Half-life (t1/2) of Padsevonil During Part B
Description: t1/2 is the apparent terminal half-life of padsevonil.
Time Frame: Predose up to 12 hours postdose
Population: as for outcome 3
Arm/Group | Part B: PSL
Number analyzed (Participants) | 0

12. Secondary Outcome: Half-life (t1/2) of Cannabidiol During Part B
Description: t1/2 is the apparent terminal half-life of CBD.
Time Frame: Predose up to 12 hours postdose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Part B: CBD (PKS)
Number analyzed (Participants) | 16
hours | NA [NA to NA] — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

13. Secondary Outcome: Apparent Total Body Clearance at Steady State (CLss/F) of Padsevonil During Part B
Description: CLss/F is the apparent total body clearance at steady state following extravascular administration of padsevonil.
Time Frame: Predose up to 12 hours postdose
Population: as for outcome 3
Arm/Group | Part B: PSL
Number analyzed (Participants) | 0

14. Secondary Outcome: Apparent Total Body Clearance at Steady State (CLss/F) of Cannabidiol During Part B
Description: CLss/F is the apparent total body clearance at steady state following extravascular administration of CBD.
Time Frame: Predose up to 12 hours postdose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: liter per hour
Arm/Group | Part B: CBD (PKS)
Number analyzed (Participants) | 16
liter per hour | NA [NA to NA] — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

15. Secondary Outcome: Percentage of Smooth Pursuit Eye Movements During Part B
Description: Smooth pursuit to assess eye movement coordination and attention to evaluate the ethanol effect. The average percentage of smooth pursuit for all stimulus frequencies was used as a parameter.
Time Frame: Treatment Period 1: Screening, Day 1 and Day 2
Population: FAS consisted of all study participants that were randomized, received study medication, and had at least one valid post-baseline primary pharmacodynamic assessment observation.
Measure: Mean (Standard Deviation); unit: percentage of eye movements
Groups:
- Part B: CBD (FAS): Participants received a single oral dose of CBD 10 mg/kg solution, under fasted condition on Day 1 during TP1. Participants formed the FAS.
Arm/Group | Part B: CBD (FAS)
Number analyzed (Participants) | 16
percentage of eye movements | NA (NA) — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

16. Secondary Outcome: Saccadic Peak Velocity to Assess Sedation on Day 1 of Period 1 or Day 3 of Period 2 During Part A
Description: Sixteen saccades were recorded with interstimulus intervals varying randomly. Average values of latency (reaction time), saccadic peak velocity of all correct saccades, and inaccuracy of all saccades were used as parameters. Participants received either ethanol or placebo on Day 1 of Period 1 or on Day 3 of Period 2. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours postdose on Day 1 of Period 1 or Day 3 of Period 2
Population: FAS consisted of all study participants that were randomized, received study medication, and had at least one valid post-baseline primary pharmacodynamic assessment observation. Here, n (number analyzed) signifies participants evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | Part A: Ethanol (FAS) | Part A: Placebo (FAS)
Number analyzed (Participants) | 24 | 23
degrees per second
  Predose | 497.873 (36.988) | 502.917 (32.543)
  0.5 hour: number analyzed (Participants) | 23 | 22
  0.5 hour | 471.465 (37.890) | 502.427 (47.354)
  1 hour: number analyzed (Participants) | 23 | 23
  1 hour | 458.726 (34.284) | 488.761 (35.226)
  2 hours | 455.138 (34.045) | 484.243 (37.299)
  3 hours: number analyzed (Participants) | 22 | 23
  3 hours | 455.445 (43.890) | 479.852 (33.906)
  4 hours: number analyzed (Participants) | 22 | 21
  4 hours | 459.700 (54.621) | 468.029 (36.669)
  5 hours: number analyzed (Participants) | 23 | 23
  5 hours | 447.909 (29.508) | 484.778 (32.631)
  6 hours: number analyzed (Participants) | 23 | 22
  6 hours | 466.417 (37.985) | 479.150 (37.994)
  8 hours: number analyzed (Participants) | 23 | 23
  8 hours | 474.283 (33.625) | 486.883 (38.078)
  10 hours: number analyzed (Participants) | 23 | 22
  10 hours | 484.513 (33.232) | 489.495 (38.495)

17. Secondary Outcome: Saccadic Peak Velocity to Assess Sedation on Day 5 of Period 4 or Day 7 of Period 5 During Part A
Description: Sixteen saccades were recorded with interstimulus intervals varying randomly. Average values of latency (reaction time), saccadic peak velocity of all correct saccades, and inaccuracy of all saccades were used as parameters. Participants received either ethanol or placebo on Day 5 of Period 4 or Day 7 of Period 5. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours postdose on Day 5 of Period 4 or Day 7 of Period 5
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | Part A: PSL + Ethanol (FAS) | Part A: PSL + Placebo (FAS)
Number analyzed (Participants) | 23 | 23
degrees per second
  Predose: number analyzed (Participants) | 23 | 22
  Predose | 481.335 (40.894) | 466.509 (43.334)
  0.5 hour: number analyzed (Participants) | 23 | 20
  0.5 hour | 434.465 (48.160) | 454.980 (35.882)
  1 hour: number analyzed (Participants) | 23 | 22
  1 hour | 405.517 (50.706) | 427.505 (42.232)
  2 hours: number analyzed (Participants) | 22 | 21
  2 hours | 414.268 (61.752) | 418.748 (49.071)
  3 hours: number analyzed (Participants) | 21 | 21
  3 hours | 401.548 (46.004) | 423.543 (51.720)
  4 hours: number analyzed (Participants) | 21 | 21
  4 hours | 410.386 (47.324) | 442.152 (46.641)
  5 hours: number analyzed (Participants) | 21 | 21
  5 hours | 418.252 (41.277) | 450.319 (38.954)
  6 hours: number analyzed (Participants) | 22 | 21
  6 hours | 436.268 (55.152) | 470.576 (47.370)
  8 hours: number analyzed (Participants) | 23 | 21
  8 hours | 480.891 (41.106) | 467.162 (37.902)
  10 hours: number analyzed (Participants) | 22 | 21
  10 hours | 474.209 (41.119) | 466.933 (43.241)

18. Secondary Outcome: Saccadic Peak Velocity to Assess Sedation During Part B
Description: Sixteen saccades were recorded with interstimulus intervals varying randomly. Average values of latency (reaction time), saccadic peak velocity of all correct saccades, and inaccuracy of all saccades were used as parameters.
Time Frame: Treatment Period 1: Screening, Day 1 and Day 2
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | Part B: CBD (FAS)
Number analyzed (Participants) | 16
degrees per second | NA (NA) — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

19. Secondary Outcome: Adaptive Tracking to Assess Visuo-Motor Control and Vigilance on Day 1 of Period 1 or Day 3 of Period 2 During Part A
Description: The adaptive tracking test was performed as originally described by Borland and Nicholson (Borland and Nicholson, 1984). Performance was scored after a fixed period of 3.5 minutes and reflected visuo-motor control and vigilance. The average performance scores were used in the analysis. Participants received either ethanol or placebo on Day 1 of Period 1 or on Day 3 of Period 2. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours postdose on Day 1 of Period 1 or Day 3 of Period 2
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percentage of time correctly tracked
Arm/Group | Part A: Ethanol (FAS) | Part A: Placebo (FAS)
Number analyzed (Participants) | 24 | 23
percentage of time correctly tracked
  Predose | 32.3704 (5.5709) | 32.0037 (5.6751)
  0.5 hour | 29.0825 (4.8924) | 32.0770 (5.7220)
  1 hour | 28.7825 (5.0093) | 32.0530 (5.6913)
  2 hours | 27.6325 (4.6875) | 32.6526 (5.5194)
  3 hours: number analyzed (Participants) | 23 | 23
  3 hours | 26.5765 (5.9118) | 32.3087 (6.0354)
  4 hours: number analyzed (Participants) | 23 | 23
  4 hours | 26.4087 (6.5784) | 31.8835 (6.0274)
  5 hours: number analyzed (Participants) | 23 | 23
  5 hours | 27.9500 (5.1829) | 32.0752 (5.8386)
  6 hours: number analyzed (Participants) | 23 | 23
  6 hours | 28.9587 (5.6291) | 32.0757 (5.6722)
  8 hours: number analyzed (Participants) | 23 | 23
  8 hours | 31.0778 (5.7553) | 32.0300 (5.8507)
  10 hours: number analyzed (Participants) | 23 | 23
  10 hours | 32.5391 (5.2327) | 33.3322 (5.9769)

20. Secondary Outcome: Adaptive Tracking to Assess Visuo-Motor Control and Vigilance on Day 5 of Period 4 or Day 7 of Period 5 During Part A
Description: The adaptive tracking test was performed as originally described by Borland and Nicholson (Borland and Nicholson, 1984). Performance was scored after a fixed period of 3.5 minutes and reflected visuo-motor control and vigilance. The average performance scores were used in the analysis. Participants received either ethanol or placebo on Day 5 of Period 4 or Day 7 of Period 5. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours on Day 5 of Period 4 or Day 7 of Period 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time correctly tracked
Arm/Group | Part A: PSL + Ethanol (FAS) | Part A: PSL + Placebo (FAS)
Number analyzed (Participants) | 23 | 22
percentage of time correctly tracked
  Predose | 30.5017 (7.0354) | 29.0691 (7.1405)
  0.5 hour | 23.3339 (6.4727) | 25.8650 (7.7624)
  1 hour | 19.4317 (7.5471) | 20.5714 (7.7253)
  2 hours | 17.1617 (6.8895) | 19.3395 (7.8659)
  3 hours | 18.4870 (6.9150) | 25.0859 (7.2415)
  4 hours | 18.8713 (7.9952) | 27.5827 (6.8106)
  5 hours | 20.4422 (8.3476) | 29.4377 (6.5829)
  6 hours | 26.3652 (6.5759) | 30.3214 (6.4549)
  8 hours | 30.3570 (6.3134) | 31.3282 (5.9957)
  10 hours | 30.6039 (6.5557) | 31.9223 (7.1749)

21. Secondary Outcome: Adaptive Tracking to Assess Visuo-Motor Control and Vigilance During Part B
Description: The adaptive tracking test was performed as originally described by Borland and Nicholson (Borland and Nicholson, 1984). Performance was scored after a fixed period of 3.5 minutes and reflected visuo-motor control and vigilance.
Time Frame: Treatment Period 1: Screening, Day 1 and Day 2
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of time correctly tracked
Arm/Group | Part B: CBD (FAS)
Number analyzed (Participants) | 16
percentage of time correctly tracked | NA (NA) — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

22. Secondary Outcome: Body Sway to Assess Postural Stability on Day 1 of Period 1 or Day 3 of Period 2 During Part A
Description: Body Sway test measured the study participant's body movements in a single direction. Body sway was measured by CHCR NeuroCart. Study participants were asked to stand erect and motionless with their eyes closed. The amplitude and direction of any Body Sway was recorded for 1 minute. Participants received either ethanol or placebo on Day 1 of Period 1 or on Day 3 of Period 2. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours postdose on Day 1 of Period 1 or Day 3 of Period 2
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Part A: Ethanol (FAS) | Part A: Placebo (FAS)
Number analyzed (Participants) | 24 | 23
millimeters
  Predose | 234.258 (131.198) | 219.348 (123.362)
  0.5 hour | 390.671 (293.387) | 238.083 (108.227)
  1 hour | 379.246 (226.889) | 235.613 (115.707)
  2 hours | 410.292 (307.000) | 258.348 (133.061)
  3 hours: number analyzed (Participants) | 23 | 23
  3 hours | 392.813 (300.259) | 251.109 (141.894)
  4 hours: number analyzed (Participants) | 23 | 23
  4 hours | 410.500 (277.375) | 241.361 (123.019)
  5 hours: number analyzed (Participants) | 23 | 23
  5 hours | 380.043 (238.041) | 240.322 (131.546)
  6 hours: number analyzed (Participants) | 22 | 23
  6 hours | 298.445 (177.888) | 285.191 (193.643)
  8 hours: number analyzed (Participants) | 23 | 23
  8 hours | 254.830 (134.773) | 252.930 (166.126)
  10 hours: number analyzed (Participants) | 23 | 23
  10 hours | 244.057 (146.336) | 239.283 (138.579)

23. Secondary Outcome: Body Sway to Assess Postural Stability on Day 5 of Period 4 or Day 7 of Period 5 During Part A
Description: Body Sway test measured the study participant's body movements in a single direction. Body sway was measured by CHCR NeuroCart. Study participants were asked to stand erect and motionless with their eyes closed. The amplitude and direction of any Body Sway was recorded for 1 minute. Participants received either ethanol or placebo on Day 5 of Period 4 or Day 7 of Period 5. Therefore, the results were summarized by treatment.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8 and 10 hours on Day 5 of Period 4 or Day 7 of Period 5
Population: FAS consisted of all study participants that were randomized, received study medication, and had at least one valid post-baseline primary pharmacodynamic assessment observation. Here, Number of participants analyzed signifies participants who were evaluable for the assessment and n (number analyzed) signifies participants evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Part A: PSL + Ethanol (FAS) | Part A: PSL + Placebo (FAS)
Number analyzed (Participants) | 23 | 22
millimeters
  Predose | 294.843 (227.524) | 317.484 (321.623)
  0.5 hour | 746.161 (648.448) | 661.550 (943.498)
  1 hour | 1091.639 (965.116) | 863.255 (986.913)
  2 hours | 1170.452 (1118.424) | 712.391 (646.223)
  3 hours: number analyzed (Participants) | 22 | 22
  3 hours | 924.800 (873.486) | 499.077 (353.668)
  4 hours | 903.100 (888.205) | 406.586 (279.517)
  5 hours | 666.987 (735.498) | 353.905 (277.036)
  6 hours | 489.261 (431.766) | 335.400 (256.120)
  8 hours | 314.713 (242.121) | 277.614 (189.464)
  10 hours | 274.696 (180.248) | 247.100 (137.795)

24. Secondary Outcome: Body Sway to Assess Postural Stability During Part B
Description: Body Sway test measured the study participant's body movements in a single direction. Body sway was measured by CHCR NeuroCart. Study participants were asked to stand erect and motionless with their eyes closed. The amplitude and direction of any Body Sway was recorded for 1 minute.
Time Frame: Treatment Period 1: Screening, Day 1 and Day 2
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Part B: CBD (FAS)
Number analyzed (Participants) | 16
millimeters | NA (NA) — Analysis of this outcome measure was not performed because the study was terminated. At that time, Part A had been completed, and 16 study participants had been treated with CBD in Treatment Period 1 of Part B.

25. Secondary Outcome: Number of Participants With Adverse Events During Part A
Description: An adverse event (AE) was any untoward medical occurrence in a participant or trial participant that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Screening up to the Safety Follow-up visit of Part A (up to Day 26)
Population: Safety Set consisted of all study participants who were randomized and had received at least 1 dose (any amount) of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Pre-treatment (SS): Participants with adverse events with a start date prior to the first dose of treatment were summarized in this group for Part A. Participants formed SS.
- Part A: Placebo (SS): Participants received matching placebo (for ethanol IV infusion) on Day 1 during TP1 in Treatment Sequence A and B and on Day 1 during TP2 in Treatment Sequence C and D. Participants formed the Safety Set (SS).
- Part A: Ethanol (SS): Participants received ethanol 0.6 g/L IV infusion on Day 1 during TP1 in Treatment Sequence A and B and on Day 1 during TP2 in Treatment Sequence C and D. Participants formed the SS.
- Part A: PSL (SS): Participants received PSL 100 mg or 200 mg oral tablets BID on Day 1 to 4 during TP3 in Treatment Sequence A, B, C and D. Participants formed the SS.
- Part A: PSL + Ethanol (SS): Participants received PSL 200 mg BID oral tablets + Ethanol IV infusion on Day 5 during TP4 in Treatment Sequence A and C and on Day 7 during TP5 in Treatment Sequence B and D. Participants formed the SS.
- Part A: PSL + Placebo (SS): Participants received PSL oral tablets 100 mg or 200 mg + Placebo (for ethanol IV infusion) on Day 7 during TP5 in Treatment Sequence A and C and on Day 5 during TP4 in Treatment Sequence B and D. Participants formed the SS.
Arm/Group | Part A: Pre-treatment (SS) | Part A: Placebo (SS) | Part A: Ethanol (SS) | Part A: PSL (SS) | Part A: PSL + Ethanol (SS) | Part A: PSL + Placebo (SS)
Number analyzed (Participants) | 24 | 23 | 24 | 23 | 23 | 23
Participants | 8 | 6 | 17 | 22 | 22 | 20

26. Secondary Outcome: Number of Participants With Adverse Events During Part B
Description: An AE was any untoward medical occurrence in a participant or trial participant that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Screening up to the Safety Follow-up visit of Part B (up to Day 66)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Pre-treatment (SS): Participants with adverse events with a start date prior to the first dose of treatment were summarized in this group for Part B. Participants formed SS.
- Part B: CBD (SS): Participants received a single oral dose of CBD 10 mg/kg solution, under fasted condition on Day 1 during TP1. Participants formed the SS.
Arm/Group | Part B: Pre-treatment (SS) | Part B: CBD (SS)
Number analyzed (Participants) | 16 | 16
Participants | 2 | 11

27. Secondary Outcome: Number of Participants With Serious Adverse Events During Part A
Description: A serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, is life-threatening, required in patient hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect, is an infection that requires treatment parenteral antibiotics, other important medical events which based on medical or scientific judgement may jeopardize the participants, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Screening up to the Safety Follow-up visit of Part A (up to Day 26)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pre-treatment (SS) | Part A: Placebo (SS) | Part A: Ethanol (SS) | Part A: PSL (SS) | Part A: PSL + Ethanol (SS) | Part A: PSL + Placebo (SS)
Number analyzed (Participants) | 24 | 23 | 24 | 23 | 23 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Number of Participants With Serious Adverse Events During Part B
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, is life-threatening, required in patient hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect, is an infection that requires treatment parenteral antibiotics, other important medical events which based on medical or scientific judgement may jeopardize the participants, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Screening up to the Safety Follow-up visit of Part B (up to Day 66)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Pre-treatment (SS) | Part B: CBD (SS)
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

29. Secondary Outcome: Number of Participants With Treatment-related Adverse Events During Part A
Description: Treatment-related adverse event was an adverse event for which a causal relationship between the product and the occurrence is suspected.
Time Frame: From Baseline up to Safety Follow-up visit of Part A (up to Day 26)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo (SS) | Part A: Ethanol (SS) | Part A: PSL (SS) | Part A: PSL + Ethanol (SS) | Part A: PSL + Placebo (SS)
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 23
Participants | 1 | 5 | 21 | 20 | 18

30. Secondary Outcome: Number of Participants With Treatment-related Adverse Events During Part B
Description: as for outcome 29
Time Frame: From Baseline up to Safety Follow-up visit of Part B (up to Day 66)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: CBD (SS)
Number analyzed (Participants) | 16
Participants | 7

31. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation of the Study During Part A
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Screening up to Safety Follow-up visit of Part A (up to Day 26)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pre-treatment (SS) | Part A: Placebo (SS) | Part A: Ethanol (SS) | Part A: PSL (SS) | Part A: PSL + Ethanol (SS) | Part A: PSL + Placebo (SS)
Number analyzed (Participants) | 24 | 23 | 24 | 23 | 23 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation of the Study During Part B
Description: as for outcome 31
Time Frame: From Screening up to Safety Follow-up visit of Part B (up to Day 66)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Pre-treatment (SS) | Part B: CBD (SS)
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Screening up to Safety Follow-up visit of Part A (up to Day 26) and of Part B (up to Day 66)
Description: An AE was any untoward medical occurrence in a participant or trial participant that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
Arm/Group | Part A: Pre-treatment (SS) | Part A: Placebo (SS) | Part A: Ethanol (SS) | Part A: PSL (SS) | Part A: PSL + Ethanol (SS) | Part A: PSL + Placebo (SS) | Part B: Pre-treatment (SS) | Part B: CBD (SS)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/24 | 0/23 | 0/23 | 0/23 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/24 | 0/23 | 0/23 | 0/23 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/24 | 4/23 | 17/24 | 22/23 | 22/23 | 18/23 | 2/16 | 11/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pre-treatment (SS) (N=24) | Part A: Placebo (SS) (N=23) | Part A: Ethanol (SS) (N=24) | Part A: PSL (SS) (N=23) | Part A: PSL + Ethanol (SS) (N=23) | Part A: PSL + Placebo (SS) (N=23) | Part B: Pre-treatment (SS) (N=16) | Part B: CBD (SS) (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 8 (8) | 2 (3) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2) | 9 (11) | 3 (4) | 2 (2) | 0 (0) | 2 (2)
Feeling Drunk (General disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 1 (1) | 9 (9) | 0 (0) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anterograde amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 6 (7) | 17 (30) | 7 (7) | 1 (1) | 0 (0) | 2 (2)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5) | 7 (13) | 7 (10) | 1 (1) | 2 (2) | 3 (3)
Slow response to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 20 (43) | 15 (23) | 14 (26) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden onset of sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (33) | 6 (9) | 3 (3) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Illusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Negative thoughts (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated because the decision was made to terminate the PSL development program in focal-onset seizures on 22 May 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT04039919/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT04039919/SAP_001.pdf